CLINICAL TRIAL: NCT04456439
Title: Intermediate-size Expanded Access of Remestemcel-L, Human Mesenchymal Stromal Cells, for Multisystem Inflammatory Syndrome in Children (MIS-C) Associated With Coronavirus Disease (COVID-19)
Brief Title: Intermediate-size Expanded Access Program (EAP), Mesenchymal Stromal Cells (MSC) for Multisystem Inflammatory Syndrome in Children (MIS-C) Associated With Coronavirus Disease (COVID-19)
Status: No longer available | Type: Expanded Access
Sponsor: Mesoblast International Sàrl (Industry)
Responsible Party: Sponsor
Organization: Mesoblast, Ltd. (Industry)
Other Study IDs: MSB-MSC-MISC001
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Multisystem Inflammatory Syndrome in Children (MIS-C) Associated With Coronavirus Disease (COVID-19)
Keywords: MIS-C; COVID-19; MSC; remestemcel-L; Mesoblast; mesenchymal; cellular therapy; cells
MeSH Terms: conditions — pediatric multisystem inflammatory disease, COVID-19 related; COVID-19 | interventions — remestemcel-l; Hydrocortisone; Diphenhydramine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Biological: Remestemcel-L — Participants may receive up to 2 infusions of 2 x 10^6 remestemcel-L within a 5-day period.
Drug: Hydrocortisone — Participants who are not currently taking a corticosteroid will receive hydrocortisone, 0.5-1 milligram per kilogram (mg/kg), up to 50 mg IV, at least 30 minutes prior to the infusion of remestemcel-L.
Drug: Diphenhydramine — Participants will receive diphenhydramine, 0.5-1 mg/kg, up to 50 mg IV, at least 30 minutes prior to the infusion of remestemcel-L.
  Other Names: Benadryl®

SUMMARY:
The objectives of this intermediate-size expanded access protocol are to assess the safety and efficacy of remestemcel-L in participants with MIS-C associated with COVID-19.

DETAILED DESCRIPTION:
This intermediate-size expanded access protocol plans to treat approximately 50 children or adolescents, male and female, with MIS-C associated with COVID-19. Participants who are 2 months to 17 years of age, inclusive, will be enrolled at multiple clinical sites across the United States.

ELIGIBILITY:
Inclusion Criteria

1. 2 months to 17 years of age, inclusive
2. Positive for current or recent SARS-CoV-2 (COVID-19) infection by real-time reverse transcription polymerase chain reaction (RT-PCR), serology, or antigen test; or COVID-19 exposure within the 4 weeks prior to the onset of symptoms AND no alternative plausible diagnoses
3. Presenting with:

   * Fever (>38.0°C or >100.4°F for ≥24 hours) or reporting subjective fever lasting ≥24 hours
   * Laboratory evidence of inflammation with high sensitivity C-reactive protein (hsCRP) ≥4.0 milligrams per deciliter (mg/dL) and associated abnormalities of at least one of the following:

     * elevated erythrocyte sedimentation rate (ESR)
     * elevated fibrinogen
     * elevated procalcitonin
     * elevated d-dimer
     * elevated ferritin
     * elevated lactic dehydrogenase (LDH)
     * elevated interleukin 6 (IL-6)
     * elevated neutrophils
     * reduced lymphocytes
     * low albumin
   * Clinically severe multisystem illness requiring hospitalization with evidence for cardiac involvement plus at least one other organ involvement (renal, respiratory, hematologic, gastrointestinal, dermatologic or neurological)

     * Cardiac involvement is defined as reduced left ventricular ejection fraction (<55%) in addition to at least one of the following:

       * increased troponin I,
       * increased N-terminal pro-B-type natriuretic peptide (NT-proBNP) or BNP and/or
       * echocardiographic and/or other imaging evidence of left anterior descending coronary artery (LAD) and/or right coronary artery (RCA) dilation associated with a z-score > 2.5
4. If on mechanical ventilation or ECMO, ≤72 hours post initiation of the respiratory support device

Exclusion Criteria

1. Documented other microbial cause for MIS-C including bacterial sepsis, staphylococcal or streptococcal shock syndromes, or infections associated with myocarditis such as enterovirus. Of importance, waiting for results of these investigations should not delay initiation of remestemcel-L therapy.
2. Females who are pregnant or lactating
3. Body mass index (BMI) ≥40 kilograms per square meter (kg/m^2)
4. Known hypersensitivity to dimethyl sulfoxide (DMSO) or to porcine or bovine proteins
5. Aspartate aminotransferase/alanine transaminase (AST/ALT) ≥5x upper limit of normal (ULN)
6. Creatinine clearance <30 mL/min
7. Serum creatinine >2 mg/dL
8. Any end-stage organ disease which in the opinion of the treating physician may possibly affect the safety of the remestemcel-L treatment.

Ages: 2 Months to 17 Years | Sex: All
Age Groups: Child

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth M. Borow, MD, Study Director — Mesoblast, Inc.

REFERENCES:
- [Result] Eckard AR, Borow KM, Mack EH, Burke E, Atz AM. Remestemcel-L Therapy for COVID-19-Associated Multisystem Inflammatory Syndrome in Children. Pediatrics. 2021 May;147(5):e2020046573. doi: 10.1542/peds.2020-046573. Epub 2021 Feb 12. PMID 33579813